CLINICAL TRIAL: NCT06070311
Title: Effect of Thymoquinone and Olive Oil on Wound Healing After Endoscopic Sinus Surgery in Patients With Nasal Polyposis
Brief Title: Wound Healing After Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tarek Ashraf Abdelhasib, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: endoscopic sinus surgery
Record Dates: First submitted 2023-09-21; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Nasal Polyps; Chronic Sinusitis
MeSH Terms: conditions — Nasal Polyps | interventions — thymoquinone

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thymoquinone (0.5%) and Olive oil ointment (Active Comparator): thymoquinone (0.5%) and olive oil ointment will be applied to fill the ethmoidal and different sinuses cavities of one randomly chosen side of the nose.
  Interventions: Combination Product: Thymoquinone (0.5%) and Olive oil ointment
- No intervention (No Intervention): no intervention

INTERVENTIONS:
Combination Product: Thymoquinone (0.5%) and Olive oil ointment — Preparation of the Thymoquinone and Olive oil ointment:
  Thymoquinone Oleaginous base ointment containing olive oil will be prepared for intranasal administration. The ointment will be prepared using the fusion method as follows:
  Anhydrous lanolin and white soft paraffin will be melted at 70°C and then olive oil will be added with continuous stirring, Thymoquinone will be added to the congealing mixture as it is being cooled and stirred finally, the congealing mixture is left to cool at room temperature tell solidification and sterilized using UV radiation. The final product will be characterized for spreadability, drug content, drug release and stability.
  Other Names: thymoquinone and olive oil ointment
  Arms: Thymoquinone (0.5%) and Olive oil ointment

SUMMARY:
This study aims to determine the effect of Thymoquinone (0.5%) and olive oil ointment on Wound healing after Endoscopic sinus surgery.

DETAILED DESCRIPTION:
Endoscopic sinus surgery (ESS) has become a widely accepted procedure for medically refractory chronic rhino sinusitis and nasal polyps. Over 250,000 endoscopic sinus surgeries are performed yearly in the United States alone, however, postoperative complications and disease recurrence requiring revision surgery are reported in 14% to 24% of patients in long-term follow-up.

There is an increasing interest in interventions and therapies targeted at optimizing outcomes and preventing revision surgery which often depends on good wound healing and less adhesion formation.

The choice of appropriate post-surgical topical treatments is important for healing time and for preventing mucosal complications such as adhesions, crusting formation, and atrophy with secondary bacterial and fungal infections in this light this study aims to determine the effect of thymoquinone and olive oil ointment on wound healing after ESS.

Thymoquinone (TQ) is the most abundant constituent of the volatile oil of Nigella sativa seeds and most properties of Nigella sativa are mainly attributed to TQ. Several pharmacological actions and therapeutic potentials of TQ have been investigated including being antioxidant, anti-inflammatory, antihistaminic, antimicrobial, anti-allergic, anti-fibrotic, and anti-cancer.

Olive oil plays an important role in wound healing process due to its content of phenolic compounds accelerating wound healing through their anti-inflammatory, antioxidant, and antimicrobial properties and their stimulation of angiogenic activities required for granulation tissue formation and wound re-epithelialization.

This Double Blinded Randomized Prospective Comparative study will follow patients with nasal polyposis who are indicated for endoscopic sinus surgery at the Department of Otorhinolaryngology in Assiut University Hospital during the period from the 1st of October 2023 to the 31st of September 2025.

At baseline (before surgery), a full medical history, an otorhinolaryngological examination, and pre-operative screening will be performed to ensure eligibility for the study. The patients will be informed about the surgical procedures, the potential risks of the surgery, and the aim and methodology of the study.

(A) Preoperative:

Full history taking:

1. Personal History
2. History of Sino-nasal symptoms e.g., nasal obstruction, nasal discharge, headache, hyposmia, facial congestion, etc.
3. Other ENT symptoms
4. General symptoms e.g., asthma, allergy, etc.
5. Medical history e.g., steroids, antibiotics, anticholinergics, etc.
6. History of nasal surgery
7. SNOT 22 questionnaire: To assess preoperative severity of symptoms.

Full medical examination:

1. General examination
2. Full ENT examination
3. Nasal Endoscopy:

   * To evaluate polyp size, site, extent, and consistency.

Investigations:

1. Routine preoperative investigations: CBC, prothrombin time and concentration
2. Radiological investigations: Multi-slice CT scan of the nose and paranasal sinuses axial and coronal cuts without contrast and each patient will be scored according to Lund-Mackay CT scoring.

Preparation of the Thymoquinone and Olive oil ointment:

Thymoquinone Oleaginous base ointment containing olive oil will be prepared for intranasal administration. The ointment will be prepared using the fusion method as follows:

Anhydrous lanolin and white soft paraffin will be melted at 70°C and then olive oil will be added with continuous stirring, Thymoquinone will be added to the congealing mixture as it is being cooled and stirred finally, the congealing mixture is left to cool at room temperature tell solidification and sterilized using UV radiation. The final product will be characterized for spreadability, drug content, drug release and stability.

(B) Intraoperative: All cases will be performed under general anaesthesia and the ESS procedure performed by the senior author is that defined by Kennedy.

Immediately after performing the ESS, Thymoquinone and olive oil Ointment will be applied to fill the ethmoidal and different sinuses cavities of one randomly chosen side of the nose, the selected side will be chosen randomly using the following online randomizer tool:

Randomizer | Random Name/Number Picker - AnnaBet.com Then nasal packing with nasal sponge will be done for both sides.

(C) Postoperative: Patients will attend routine follow-up at 1, 2,3,4,8 and 12 weeks after surgery. At these visits, an endoscopic inspection will be performed, and the patients will undergo debridement of the ethmoid cavities when necessary. In addition, endoscopic data regarding the health of the Sino nasal mucosa will be collected. An independent investigator blinded to the side of TQ, and olive oil ointment placement will assess and compare the wound healing in both sides regarding adhesions, crust formation, granulation, infection and score each item using the scoring mentioned below.

Crust formation:

0: No crust formation observed.

1. Thin and easily removable crusts.
2. Moderate crust formation, requiring gentle removal.
3. Thick and adherent crusts, requiring careful and meticulous removal.

Adhesions:

0: No adhesions observed.

1. Mild adhesions, limited to small areas.
2. Moderate adhesions, affecting larger areas but without complete obstruction.
3. Severe adhesions, causing significant obstruction and impaired sinus drainage. 3.Granulation:

0: No granulations observed.

1. Mild granulation tissue, with minimal vascularity and minimal elevation.
2. Moderate granulation tissue, with moderate vascularity and noticeable elevation.
3. Severe granulation tissue, with marked vascularity and significant elevation. 4.Infection:

0: No signs or symptoms of infection observed.

1. Mild infection, mucopurulent discharge limited to small area of the ethmoidal cavity.
2. Moderate infection, mucopurulent discharge filling one sinus.
3. Severe infection, mucopurulent discharge filling more than one sinus.

Participants will take the SNOT-22 questionnaire after the operation at the follow up visits to evaluate sino nasal symptoms.

ELIGIBILITY:
Inclusion Criteria:

- All patients who will be clinically diagnosed and radiologically confirmed cases with bilateral nasal polyposis indicated for Endoscopic sinus surgery.

Exclusion Criteria:

1. Unfit patient for surgery
2. Pregnant and lactating women.
3. Patients unwilling to participate.
4. Patients who have unilateral disease.
5. Patients with a history of the following underlying medical conditions, which are associated with an increased rate of revision surgery, will be excluded from the study:

   1. Aspirin intolerance
   2. Asthma
   3. Mucociliary disorder
   4. Immunocompromised status.
6. Patients with known allergic reactions to Thymoquinone or olive oil.
7. Injury of the orbit with any tear in the periorbital area.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Determining the effectiveness of Thymoquinone (0.5%) and olive oil on Wound healing after Endoscopic sinus surgery regarding crust formation by Endoscopic examination. | Patients will attend routine follow-up at 1, 2,3,4,8 and 12 weeks after surgery
  Endoscopic data regarding the health of the Sino nasal mucosa will be collected. An independent investigator blinded to the side of TQ, and olive oil ointment placement will assess and compare the wound healing in both sides. crust formation will be scored as following:
  0: No crust formation observed.
  1. Thin and easily removable crusts.
  2. Moderate crust formation, requiring gentle removal.
  3. Thick and adherent crusts, requiring careful and meticulous removal.
  0 is the lowest score meaning no crusts are formed while 3 is the highest score meaning severe crusts are formed.
Determining the effectiveness of Thymoquinone (0.5%) and olive oil on Wound healing after Endoscopic sinus surgery regarding adhesions by Endoscopic examination. | Patients will attend routine follow-up at 1, 2,3,4,8 and 12 weeks after surgery
  Endoscopic data regarding the health of the Sino nasal mucosa will be collected. An independent investigator blinded to the side of TQ, and olive oil ointment placement will assess and compare the wound healing in both sides. adhesions will be scored as following:
  0: No adhesions observed.
  1. Mild adhesions, limited to small areas.
  2. Moderate adhesions, affecting larger areas but without complete obstruction.
  3. Severe adhesions, causing significant obstruction and impaired sinus drainage.
  0 is the lowest score meaning no adhesions are formed while 3 is the highest score meaning severe adhesions are formed.
Determining the effectiveness of Thymoquinone (0.5%) and olive oil on Wound healing after Endoscopic sinus surgery regarding granulation formation by Endoscopic examination | Patients will attend routine follow-up at 1, 2,3,4,8 and 12 weeks after surgery
  Endoscopic data regarding the health of the Sino nasal mucosa will be collected. An independent investigator blinded to the side of TQ, and olive oil ointment placement will assess and compare the wound healing in both sides. Granulations will be scored as following:
  0: No granulations observed.
  1. Mild granulation tissue, with minimal vascularity and minimal elevation.
  2. Moderate granulation tissue, with moderate vascularity and noticeable elevation.
  3. Severe granulation tissue, with marked vascularity and significant elevation.
  0 is the lowest score meaning no granulation tissue is formed while 3 is the highest score meaning severe granulation tissue are formed.
Determining the effectiveness of Thymoquinone (0.5%) and olive oil on Wound healing after Endoscopic sinus surgery regarding infection by Endoscopic examination. | Patients will attend routine follow-up at 1, 2,3,4,8 and 12 weeks after surgery
  Endoscopic data regarding the health of the Sino nasal mucosa will be collected. An independent investigator blinded to the side of TQ, and olive oil ointment placement will assess and compare the wound healing in both sides. Infection will be scored as following:
  0: No signs or symptoms of infection observed.
  1. Mild infection, mucopurulent discharge limited to small area of the ethmoidal cavity.
  2. Moderate infection, mucopurulent discharge filling one sinus.
  3. Severe infection, mucopurulent discharge filling more than one sinus.
  0 is the lowest score meaning there is no infection while 3 is the highest score meaning there is severe infection.

SECONDARY OUTCOMES:
Evaluation of symptoms of CRS and NP after Endoscopic Sinus Surgery using SNOT22 questionnaire. | Patients will attend routine follow-up at 1, 2,3,4,8 and 12 weeks after surgery
  Sinonasal Outcome Test (SNOT-22) Questionnaire will be taken by each participant before and after surgery. The SNOT-22 consists of 22 questions; items 1 to 12 represent the physical problems associated with rhinosinusitis, items 13 to 18 represent the functional limitations, and items 20 to 22 represent the emotional consequences. Each question is scored by the patient from 0 (no problem) to 5 (the problem is as bad as it can be). The overall score can theoretically range from 0 to 110, with higher scores reflecting more severe quality of life impairment as subjectively reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mostafa Osman, Professor, Study Chair — Assiut University; Ahmed Gamal Sholkamy, Doctor, Study Director — Assiut University; Tarek Ashraf, Doctor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Alobid I, Anton E, Armengot M, Chao J, Colas C, del Cuvillo A, Davila I, Dordal MT, Escobar C, Fernandez-Parra B, Gras-Cabrerizo JR, Ibanez MD, Lluch M, Mateu V, Montoro J, Gili JR, Mullol J, Navarro AM, Pumarola F, Rondon C, Sanchez-Hernandez MC, Sarandeses A, Soler R, Valero AL; Rhinoconjunctivitis Committee; Spanish Society of Allergy and Clinical Immunology; Rhinology and Allergy Commission; Spanish Society of Otorhinolaryngology. SEAIC-SEORL. Consensus Document on Nasal Polyposis. POLINA Project. J Investig Allergol Clin Immunol. 2011;21 Suppl 1:1-58. No abstract available. PMID 21714471
- [Background] Hastan D, Fokkens WJ, Bachert C, Newson RB, Bislimovska J, Bockelbrink A, Bousquet PJ, Brozek G, Bruno A, Dahlen SE, Forsberg B, Gunnbjornsdottir M, Kasper L, Kramer U, Kowalski ML, Lange B, Lundback B, Salagean E, Todo-Bom A, Tomassen P, Toskala E, van Drunen CM, Bousquet J, Zuberbier T, Jarvis D, Burney P. Chronic rhinosinusitis in Europe--an underestimated disease. A GA(2)LEN study. Allergy. 2011 Sep;66(9):1216-23. doi: 10.1111/j.1398-9995.2011.02646.x. Epub 2011 May 24. PMID 21605125
- [Background] Stevens WW, Schleimer RP, Kern RC. Chronic Rhinosinusitis with Nasal Polyps. J Allergy Clin Immunol Pract. 2016 Jul-Aug;4(4):565-72. doi: 10.1016/j.jaip.2016.04.012. PMID 27393770
- [Background] Bachert C, Bhattacharyya N, Desrosiers M, Khan AH. Burden of Disease in Chronic Rhinosinusitis with Nasal Polyps. J Asthma Allergy. 2021 Feb 11;14:127-134. doi: 10.2147/JAA.S290424. eCollection 2021. PMID 33603409
- [Background] Sari H, Karaketir S, Kumral TL, Akgun MF, Gurpinar B, Hanci D, Berkiten G, Uyar Y. The effect of platelet-rich fibrin (PRF) on wound healing, adhesion, and hemostasis after endoscopic sinus surgery in patients with nasal polyposis. Am J Otolaryngol. 2021 Sep-Oct;42(5):103010. doi: 10.1016/j.amjoto.2021.103010. Epub 2021 Mar 29. PMID 33862565
- [Background] Soler ZM, Smith TL. Endoscopic sinus surgery checklist. Laryngoscope. 2012 Jan;122(1):137-9. doi: 10.1002/lary.22430. Epub 2011 Nov 17. PMID 22095309
- [Background] Loftus CA, Soler ZM, Koochakzadeh S, Desiato VM, Yoo F, Nguyen SA, Schlosser RJ. Revision surgery rates in chronic rhinosinusitis with nasal polyps: meta-analysis of risk factors. Int Forum Allergy Rhinol. 2020 Feb;10(2):199-207. doi: 10.1002/alr.22487. Epub 2019 Nov 21. PMID 31752051
- [Background] Testa D, Marcuccio G, Panin G, Bianco A, Tafuri D, Thyrion FZ, Nunziata M, Piombino P, Guerra G, Motta G. Nasal mucosa healing after endoscopic sinus surgery in chronic rhinosinusitis of elderly patients: role of topic alpha-tocopherol acetate. Aging Clin Exp Res. 2017 Feb;29(Suppl 1):191-195. doi: 10.1007/s40520-016-0647-x. Epub 2016 Nov 25. PMID 27888473
- [Background] Darakhshan S, Bidmeshki Pour A, Hosseinzadeh Colagar A, Sisakhtnezhad S. Thymoquinone and its therapeutic potentials. Pharmacol Res. 2015 May-Jun;95-96:138-58. doi: 10.1016/j.phrs.2015.03.011. Epub 2015 Mar 28. PMID 25829334
- [Background] Melguizo-Rodriguez L, de Luna-Bertos E, Ramos-Torrecillas J, Illescas-Montesa R, Costela-Ruiz VJ, Garcia-Martinez O. Potential Effects of Phenolic Compounds That Can Be Found in Olive Oil on Wound Healing. Foods. 2021 Jul 15;10(7):1642. doi: 10.3390/foods10071642. PMID 34359512
- [Background] Hopkins C, Browne JP, Slack R, Lund V, Brown P. The Lund-Mackay staging system for chronic rhinosinusitis: how is it used and what does it predict? Otolaryngol Head Neck Surg. 2007 Oct;137(4):555-61. doi: 10.1016/j.otohns.2007.02.004. PMID 17903570
- [Background] Kennedy DW. Functional endoscopic sinus surgery. Technique. Arch Otolaryngol. 1985 Oct;111(10):643-9. doi: 10.1001/archotol.1985.00800120037003. PMID 4038136